CLINICAL TRIAL: NCT07346157
Title: PNOC044: Liothyronine (L-T3) in Combination With Bevacizumab, Irinotecan and Temozolomide (BIT) for Progressive or Relapsed Medulloblastoma (Cohort 1) or as Monotherapy for Medulloblastoma With Minimal Residual Disease (Cohort 2)
Brief Title: Liothyronine in Combination With BIT Regimen for Medulloblastoma With or Without Minimal Residual Disease
Acronym: PNOC044
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sabine Mueller, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Sabine Mueller, MD, PhD, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 250812; NCI-2025-08554 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2026-01-14; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Medulloblastoma; Medulloblastoma, Childhood; Medulloblastoma Recurrent
MeSH Terms: conditions — Medulloblastoma | interventions — Triiodothyronine; Bevacizumab; Vascular Endothelial Growth Factor A; Irinotecan; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1 Cohort (Cohort 1) (Experimental): Participants will be treated with a backbone of BIT. L-T3 will be administered on day 1 of each cycle at planned dose levels (DL). Once the Recommended Phase 2 Dose (RP2D) is established with dosing days 1-7, an additional cohort of 6 participants will be treated at the maximum tolerated DL for 14 days of the cycle, Dose level escalation (DLE), which, if tolerated, will become the RP2D. If DLE is not tolerated, the RP2D will become the highest tolerated DL from the prior cohort.
  Interventions: Drug: Liothyronine (L-T3); Drug: Bevacizumab; Drug: Irinotecan; Drug: Temozolomide (TMZ)
- Phase 2 Cohort 1- Relapsed/Progressive Disease (Experimental): Participants will be treated at the RP2D of L-T3 based on the results of the safety Phase 1 cohort. Participants may continue therapy for up to 12 cycles if there is no evidence of unacceptable toxicity, disease progression, or withdrawal of consent. For participants that are benefiting from therapy, they may continue L-T3 monotherapy for one additional year (24 cycles total therapy). Treatment beyond that specified in the protocol should be discussed with the study chairs. Duration of Follow up Participants will enter follow up after the 30-day toxicity period.
  Follow-up procedures are to be captured under the PNOC COMP protocol with the exception of protocol defined follow up procedures. Participants will be followed under the PNOC COMP protocol until death or withdrawal from study.
  Interventions: Drug: Liothyronine (L-T3); Drug: Bevacizumab; Drug: Irinotecan; Drug: Temozolomide (TMZ)
- Phase 2 Cohort 2 - cfDNA positive in CSF (Experimental): Children and young adults with medulloblastoma and CSF cf-DNA positivity without radiographic disease progression/recurrence following standard upfront therapy. will include children and young adults with medulloblastoma and positive cf-DNA in CSF following initial standard therapy and will involve a Phase 2 to evaluate clearance of cf-DNA positive disease in CSF in response to L-T3 monotherapy at the RP2D. Cohort 2 will begin enrolling once the RP2D of L-T3 is established.
  Interventions: Drug: Liothyronine (L-T3)

INTERVENTIONS:
Drug: Liothyronine (L-T3) — Given orally (PO)
  Other Names: L-T3
Drug: Bevacizumab — Given IV
  Other Names: vascular endothelial growth factor (VEGF) inhibitor; VEGF inhibitor
  Arms: Phase 1 Cohort (Cohort 1); Phase 2 Cohort 1- Relapsed/Progressive Disease
Drug: Irinotecan — Given IV
  Other Names: Camptosar
  Arms: Phase 1 Cohort (Cohort 1); Phase 2 Cohort 1- Relapsed/Progressive Disease
Drug: Temozolomide (TMZ) — Given PO
  Other Names: TMZ
  Arms: Phase 1 Cohort (Cohort 1); Phase 2 Cohort 1- Relapsed/Progressive Disease

SUMMARY:
This is a Phase 1/Phase 2 study assessing liothyronine (L-T3) immunotherapy and in combination with standard chemotherapy (bevacizumab, irinotecan and temozolomide (BIT)) in children and young adults with medulloblastoma that is relapsed or progressive after standard upfront therapy.

DETAILED DESCRIPTION:
OUTLINE: This is an intra-patient dose escalation (Phase 1 (Cohort 1)) followed by a Phase 2 (Cohort 2) study.

Cohort 1: Children and young adults with relapsed or progressive disease following standard upfront therapy (including craniospinal radiation or high dose chemotherapy with autologous stem cell rescue). evaluating the safety and efficacy of combination L-T3 with BIT. Cohort 2: Children and young adults with medulloblastoma and CSF cell-free deoxyribonucleic acid (cf-DNA) positivity without radiographic disease progression/recurrence following standard upfront therapy. This is a Phase 2 study to evaluate clearance of Circulating free DNA (cfDNA) positive disease in CSF in response to L-T3 monotherapy at the RP2D (established as part of Cohort 1; Phase 1) as single agent.

Participants may continue therapy for up to 12 cycles if there is no evidence of unacceptable toxicity, disease progression, or withdrawal of consent. For participants that are benefiting from therapy, they may continue L-T3 monotherapy for one additional year (24 cycles total therapy). Treatment beyond that specified in the protocol should be discussed with the study chairs. Duration of Follow up Participants will enter follow up after the 30-day toxicity period.

Follow-up procedures are to be captured under the Pediatric NeuroOncology Consortium (PNOC) COMP protocol with the exception of protocol defined follow up procedures. Participants will be followed under the PNOC COMP protocol until death or withdrawal from study.

The study will complete enrollment within 5 years from the time the study opens to accrual (including 3 years for enrollment and 2 years of long term follow up).

ELIGIBILITY:
Inclusion Criteria:

1. Phase 1 and Phase 2, Cohort 1:

   Participants must have histologically confirmed medulloblastoma that is relapsed/progressive following standard upfront therapy. Tissue confirmation of medulloblastoma diagnosis is required at diagnosis and not required at the time of relapse for entry into the study.
2. Phase 2, Cohort 2: Participants must have cerebrospinal fluid (CSF) with cell-free deoxyribonucleic acid (cf-DNA) + assessed in a Chemiluminescent immunoassay (CLIA)-certified or protocol-approved laboratory. After entry into the study, another CSF sample will be collected and analyzed centrally prior to initiation of protocol therapy to verify cf-DNA positivity.
3. Evidence of Disease:

   Phase 1 and Phase 2, Cohort 1:

   Participants may have either Measurable or Evaluable Disease Measurable Disease: Participants must have clear residual disease at the time of enrollment, defined as tumor that is measurable in two perpendicular dimensions on MRI Evaluable Disease: Diffuse leptomeningeal disease OR clear MRI evidence of disease that may not be measurable in two perpendicular dimensions.

   Phase 2, Cohort 2:

   For cf-DNA positive cohort: Participants are not required to have measurable or evaluable disease but must have cf-DNA positivity in a CLIA-certified or protocol-approved laboratory, as above.
4. Prior Therapy: Participants must have received standard upfront therapy for medulloblastoma (either with craniospinal radiation or high dose chemotherapy and autologous stem cell rescue. If other therapy utilized, must be discussed with study chairs prior to participation). Participants for Phase 1 and Phase 2 cohort 1 may have received further chemotherapy and/or radiation therapy beyond standard upfront therapy prior to trial enrollment. Participants within the Phase 2 cohort 1 must have experienced at least one, and at most, two relapses prior to study enrollment.
5. Age 1-25 years old.
6. Performance Score: Karnofsky ≥ 50 for participants > 16 years of age and Lansky ≥ 50 for participants ≤16 years of age (See Appendix A). Participants who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
7. For those participants currently treated with levothyroxine (Synthroid) they must have stable dosing for a minimum of 3 months prior to enrollment.
8. Organ Function Requirements

   1. Peripheral absolute neutrophil count (ANC) ≥ 1000/cubic millimeters (mm3)
   2. Platelet count ≥ 75,000/microliter (uL) (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment).
   3. A serum creatinine < 1.5 institutional/reference range upper Limit normal (ULN) based on age and gender
   4. Total bilirubin ≤ 3 x upper limit of normal (ULN); in presence of Gilbert's syndrome, total bilirubin ≤ 6 x ULN or direct bilirubin ≤ 3 x ULN

      * Alanine aminotransferase (ALT) ≤ 5 x upper limit of normal (ULN)
      * Aspartate aminotransferase (AST) ≤ 5 x ULN. 3.3.7.4 Adequate Neurologic Function Defined as:
      * Participants with seizure disorder may be enrolled if well controlled. Participants on non-enzyme inducing anticonvulsants may be excluded pending interaction(s) with study drug. 3.3.7.5 Adequate Cardiac Function Defined as:
      * Normal left ventricular systolic function on baseline transthoracic echocardiogram (TTE)
      * Normal left ventricular systolic function is defined as left ventricular ejection fraction (LVEF) >55% or shortening fraction (SF) >28%.

   AND
   * No clinically significant arrhythmia on baseline ECG (sinus arrhythmia, sinus tachycardia, sinus bradycardia, early repolarization and 1st degree atrioventricular block when partial response (PR) interval < 300 millisecond (ms) are not considered clinically significant arrhythmias).
   * In addition, the following ECG findings are not considered clinically significant in the setting of a normal echocardiogram:
   * Left axis deviation
   * Left atrial enlargement
   * Right atrial enlargement
   * Possible left ventricular hypertrophy
   * Possible right ventricular hypertrophy
   * Non-specific T wave abnormality 3.3.7.6 For the Phase 1 cohort, normal adrenal axis function is required. For those participants in the Phase 2 cohort, must have controlled adrenal insufficiency >3 months (no change in steroid replacement or stress dose plan for at least 3 months).
   * Normal adrenal axis function as defined as:
   * Morning (AM) cortisol >11mcg/deciliter (dL)
   * If AM cortisol is <11 microgram (mcg)/dL, cosyntropin stimulation test with rise to >18
9. Endocrine conditions: Participants with diabetes insipidus, diabetes melitus, or being treated with levothyroxine, must have stable dosing and control for minimum of 3 months prior to enrollment
10. For Cohort 1 only: participants must have recovered from any surgical procedure before enrolling on this study (see below for examples of major, intermediate, and minor surgical procedures):

    1. Participants with a major surgical procedure within 28 days prior to enrollment should be excluded.
    2. Participants with an intermediate surgical procedure within 14 days prior to enrollment should be excluded.
    3. For minor surgical procedures (including Broviac line or infusaport placement), participants should not receive the first planned dose of bevacizumab until the wound is healed and at least 7 days have elapsed.
    4. There should be no anticipation of need for major surgical procedures during the course of the study.
11. The effects of L-T3 with chemotherapy on the developing human fetus are unknown. For this reason and because chemotherapy agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and 4 months after completion of L-T3 and chemotherapy administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
12. Participants must be enroll on PNOC COMP if PNOC COMP is open to accrual at the enrolling institution.
13. A legal parent/guardian or participant must be able to understand, and willing to sign, a written informed consent and assent document, as appropriate.

Exclusion Criteria:

1. For Cohort 1 only: participants who have previously been treated with BIT in combination. Treatment with individual bevacizumab, irinotecan or TMZ is not an exclusion criteria.
2. Participants who have had myelosuppressive chemotherapy within 3 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier. (Participants receiving chemotherapy directly into the CSF at doses not expected to be myelosuppressive may have received therapy up to 7 days prior to enrollment).
3. Participants must be at least 7 days since the completion of therapy with a biologic or small molecule agent or non-myelosuppressive chemotherapy agent. For any agent with known adverse events that can occur beyond 7 days after administration, the period prior to enrollment must be beyond the time during which adverse events are known to occur. Such participants should also be discussed with study chairs.
4. Radiation: For participants on the Phase 1 and Phase 2 Cohort 1, the tumor designated as "measurable" for protocol purposes must not have received radiation within 6 weeks prior to study entry and focal radiation to areas of symptomatic metastatic disease must not be given within 14 days of study entry. If a new lesion occurs outside the radiation field, the participant is eligible to enroll at any time point from completion of radiation. For Cohort 2 participants, there is no required washout for radiation therapy.
5. Participants who are receiving any other investigational agents.
6. History of allergic reactions attributed to compounds of similar chemical or biologic composition to L-T3 or other agents used in study.
7. Participants receiving any medications or substances that are strong inhibitors or strong inducers of CYP450 enzymes are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently updated list such as http://medicine.iupui.edu/clinpharm/ddis/table.aspx; medical reference texts such as the Physicians' Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the participant and/or legal parent or guardian will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering.
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection.
9. Women of childbearing potential must not be pregnant or breast-feeding.
10. Human immunodeficiency virus- (HIV) positive participants will be ineligible if HIV therapy regimen has not been stable for at least 4 weeks or there is intent to change the regimen within 8 weeks following enrollment, or if they are severely immunocompromised.
11. Diagnosis of Graves' Disease or other pre-existing hyperthyroid disease.
12. Participants with severe protein calorie malnutrition that in the opinion of the investigator may not tolerate protocol therapy.
13. Participants with previous or active clinical cardiovascular disease, including the history of heart failure, myocardial infarction, cardiomyopathy, or ventricular systolic dysfunction on TTE (LVEF <55% or SF <28%), clinically significant arrhythmia (including atrial fibrillation, atrial flutter, frequent ventricular ectopy), clinically significant peripheral vascular disease.
14. Participants with uncontrolled systemic hypertension (systolic blood pressure > 95th percentile for age and height if participant is ≤ 17 years old)
15. Participants with uncontrolled diabetes mellitus (HbA1c >8%) or uncontrolled diabetes insipidus

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 69 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2031-03-31 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants experienced an Adverse Event | Up to 28 days
  Proportion of participants with adverse events of L-T3 as graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version 5.0)
Proportion of participants who experience dose-limiting toxicity (DLT) (Dose Escalation) | Up to 28 days
  The DLT evaluable analysis set includes all participants in the dose-finding part of the study who have received the target doses of L-T3, and who have either experienced a DLT or were followed for the full DLT evaluation period. DLT is defined as L-T3-related toxicity at a frequency ≥33% in any treatment arm.
Maximum Tolerated Dose (MTD) (Dose Escalation) | Up to 28 days
  The DLT evaluable analysis set includes all participants in the dose-finding part of the study who have received the target doses of L-T3, and who have either experienced a DLT or were followed for the full DLT evaluation period. The MTD is defined as the dose level given for 14 days which ≤ 1/6 participants experience a DLT.
Percentage Progressive Free Survival (PFS) at month 9 | up to 9 months
  Cohort 1 Phase 2, PFS at 9 months is defined as the proportion of patients alive and progression-free 9 months from start of treatment. Any patient lost-to-follow-up prior to 9 months will be considered an event (i.e., progression/death) for the purposes of the analysis.
Percentage of cf-DNA clearance | Up to 30 days after last dose of L-T3.
  Participants in Cohort 2 Phase 2 will be assessed in two serial measurements of at least one month apart to determine cf-DNA clearance in cerebrospinal fluid (CSF). Percentage of participants with cf-DNA clearance will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Mueller, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets will be shared with research collaborators during the course of the study.
Supporting Information: Study Protocol, SAP, ICF